CLINICAL TRIAL: NCT04708587
Title: Appropriate Duration of Anti-Platelet straTegy in Patients With Advance Chronic Kidney Disease After New Generation Drug Eluting Stents (ADAPT-CKD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2020-0073
Record Dates: First submitted 2020-12-31; First posted 2021-01-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Diseases
Keywords: anti-platelet therapy; chronic kidney disease; new generation drug eluting stents
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dual anti-platelet therapy at least 6 months (Active Comparator)
  Interventions: Drug: dual anti-platelet therapy at least 6 months
- dual anti-platelet therapy 3months or less (Experimental)
  Interventions: Drug: dual anti-platelet therapy 3months or less

INTERVENTIONS:
Drug: dual anti-platelet therapy at least 6 months — Patients enrolled in dual antiplatelets at least 6 months arm would be administered with aspirin 100mg plus clopidogrel 75mg or prasugrel 10mg once daily for at least 6 months after randomization. Clopidogrel or prasugrel should be maintained after 6 months.
  Arms: dual anti-platelet therapy at least 6 months
Drug: dual anti-platelet therapy 3months or less — Patient enrolled in the dual antiplatelet therapy less than 3 months arm would be administered with aspirin 100mg plus clopidogrel 75mg or prasugrel 10mg once daily for less than 3 months after randomization. After 3 months clopidogrel or prasugrel should be maintained.
  Arms: dual anti-platelet therapy 3months or less

SUMMARY:
The purpose of this prospective randomized clinical trial is to compare the clinical outcomes according to the duration of aspirin and clopidogrel or prasugrel with dual anti-platelet therapy after percutaneous coronary intervention in patients with advanced chronic kidney disease using a new generation drug eluting stents.

DETAILED DESCRIPTION:
Prospective, open label, multicenter randomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

1. Over 19 years old
2. Chronic Renal Failure Stage IIIb, IV, V (CKD-EPI eGFR <45 / <30 / <15 or dialysis)
3. Patients treated with a new generation drug eluting stent.
4. Patients who signed consent form

Exclusion Criteria:

1. Over 85 years old
2. Patients with high risk of bleeding 1) History of hemorrhagic stroke 2) Stroke, dementia or central nervous system damage within 1 year 3) Head trauma or brain surgery within 6 months 4) Tumor in the skull 5) If aortic dissection is suspected 6) Internal bleeding within 6 weeks 7) In case of active bleeding or bleeding disorder 8) In case of major surgery, trauma or bleeding within 3 weeks
3. Patients who need oral anticoagulant
4. Pregnant women or women of childbearing age
5. Life expectancy is less than 1 year
6. Patients with a history of intracranial bleeding
7. Moderate to severe hepatic impairment (Child-Pugh class B or C)

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2027-03-13 (Estimated); Study Completion 2028-03-13 (Estimated)

PRIMARY OUTCOMES:
Net Clinical adverse event (NACE) | 1 year
  A composite of all cause death, myocardial infarction, stent thrombosis, stroke, major bleeding (BARC 3,5)

SECONDARY OUTCOMES:
The rate of Each component of NACE | 1 year
  all cause death, myocardial infarction, stent thrombosis, stroke, major bleeding (BARC 3,5)
The rate of Cardiovascular death | 1 year
The rate of Major adverse cardiovascular events (MACE) | 1 year
  A composite of cardiovascular death, myocardial infarction, stent thrombosis or target vessel revascularization
The rate of Composite ischemic outcomes | 1 year
  A composite of cardiovascular death, myocardial infarction, stent thrombosis or ischemic stroke
The rate of major or clinically relevant nonmajor bleeding | 1 year
  BARC type 2,3,5 bleeding
Fatal bleeding | 1 year
Intracranial hemorrhage | 1 year
The rate of Target lesion revascularization | 1 year
The rate of Target vessel revascularization | 1 year
The rate of Subgroup analysis of primary endpoint, key secondary efficacy, safety endpoint and, revascularization according to the CKD stage (lllb vs. IV or V) | 1 year
The rate of Subgroup analysis of primary endpoint, key secondary efficacy, safety endpoint and, revascularization according to the clinical presentation (chronic coronary syndrome vs. acute coronary syndrome) | 1 year
he rate of Subgroup analysis of primary endpoint, key secondary efficacy, safety endpoint and, revascularization according to the type of Stent (polymer-free vs. durable-polymer) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Sun Kim, MD, PhD, FESC, Principal Investigator — Severance Hospital
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No